CLINICAL TRIAL: NCT03446599
Title: A Randomized, Placebo-controlled Single-center Pilot Study of the Hemodynamic Effects of Methylene Blue vs Hydroxocobalamin in Patients at Risk of Vasoplegia Undergoing Cardiac Surgery With Cardiopulmonary Bypass
Brief Title: Hemodynamic Effects of Methylene Blue vs Hydroxocobalamin in Patients at Risk of Vasoplegia During Cardiac Surgery
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Ying H. Low, Staff Physician, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D17173
Record Dates: First submitted 2018-02-20; First posted 2018-02-27 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Vasoplegia; Hypotension; Coronary Artery Disease; Cardiac Valve Disease
Keywords: cardiac surgery; vasoplegia; cardiopulmonary bypass
MeSH Terms: conditions — Vasoplegia; Hypotension; Coronary Artery Disease; Heart Valve Diseases | interventions — Hydroxocobalamin; Methylene Blue; Saline Solution

STUDY DESIGN:
Masking Description: Masking is unfortunately not feasible due to characteristic side effects from each medication that alert most healthcare providers to its presence: methylene blue - transient interference with pulse oximetry, blue chromaturia; hydroxocobalamin - red chromaturia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hydroxocobalamin (Experimental): Participants in this arm will receive one intravenous 5-gram dose of hydroxocobalamin reconstituted in 200ml of normal saline over 10-15minutes at the time of initiation of cardiopulmonary bypass.
  Interventions: Drug: Hydroxocobalamin
- Methyelene blue (Experimental): Participants in this arm will receive one intravenous 2mg/kg dose of methylene blue diluted in 200ml of normal saline over 10-15minutes at the time of initiation of cardiopulmonary bypass.
  Interventions: Drug: Methylene Blue
- Normal saline (Placebo Comparator): Participants in this arm will receive an intravenous administration of 200ml normal saline over 10-15minutes at the time of initiation of cardiopulmonary bypass.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Hydroxocobalamin — One intravenous dose of 5mg hydroxocobalamin, which is the current FDA-approved adult dose for carbon monoxide poisoning, reconstituted in 200ml normal saline will be administered over 10-15minutes at the time of initiation of cardiopulmonary bypass.
  Arms: Hydroxocobalamin
Drug: Methylene Blue — One intravenous dose of methylene blue 2mg/kg, which has been the accepted dose for vasoplegia, diluted in 200ml normal saline will be administered over 10-15minutes at the time of initiation of cardiopulmonary bypass.
  Arms: Methyelene blue
Drug: Normal saline — 200ml normal saline will be administered intravenously over 10-15minutes at the time of initiation of cardiopulmonary bypass.
  Arms: Normal saline

SUMMARY:
This is a pilot study to determine the hemodynamic effects when hydroxocobalamin vs methylene blue is administered during cardiopulmonary bypass in patients at risk of vasoplegia by measuring mean arterial pressure (MAP), systemic vascular resistance (SVR) and vasopressor requirement.

DETAILED DESCRIPTION:
Type of study: Randomized, placebo-controlled single-center pilot study Expected duration of subject participation: from the start of cardiac surgical procedure to 24 hours after separation from CPB.

Summary description of sequence and duration of all trial periods:

1. Recruitment and Enrollment: Patients undergoing CABG and/or valve surgery will be approached by their anesthesia provider regarding their interest in participating in this study. Those who express interest will be screened for inclusion and exclusion criteria the morning or day before scheduled surgery. Informed consent will be obtained from participants by study personnel.
2. Preoperative data will be obtained from the electronic medical record and verified with the patient: sex, age, height/weight/BSA, type of surgery, preoperative use of ACEi, beta-blocker, calcium-channel blocker, amiodarone, LVEF), and mean arterial pressure (MAP).
3. Intraoperative events, Operative and Medication Data: All participants will undergo routine induction of anesthesia. Anesthesia will be induced and maintained with midazolam, fentanyl, propofol, and isoflurane. The patient will undergo routine monitoring for all cardiac surgical patients at DHMC, which includes: arterial line mean arterial pressure (MAP, mmHg), central venous pressure (CVP, mmHg), cardiac output (CO, liters.min-1) by pulmonary artery catheter (PAC) thermodilution, serum pH, pCO2 and lactate by blood gas sampling during the pre-CPB period, during CPB and after separation from CPB, and transesophageal echocardiography (TEE). Vasopressor will be initiated and titrated to maintain MAP>60mmHg in the pre- and post-CPB period, MAP>50mmHg while on CPB, and vasopressor doses will be recorded on the anesthesia record by the providing team. After the induction of cardiopulmonary bypass, all patients will undergo non-pulsatile hypothermic (32-34 degrees celsius) CPB with a membrane oxygenator and an arterial line filter. The pump will be primed with crystalloid and serial hematocrit levels will be maintained at > 18%. Perfusion will be maintained at pump flow rates of 2-2.5L.min1.m2 throughout CPB to maintain mean arterial pressures 50-80mmg. Arterial blood gases will be measured every 20-30minutes to maintain arterial carbon dioxide partial pressures of 35-40mmHg, unadjusted for temperature (alpha-stat) and oxygen partial pressures of 150-250mmHg. An automated anesthesia record keeping system (e-DH, EPIC®™) records intraoperative hemodynamics at one-minute intervals and stores them into a networked drive. Total CPB time and cross-clamp time and intraoperative medications will also be recorded into e-DH.
4. On the initiation of CPB, participants will be randomized to: Group 1 - Hydroxocobalamin (n=20), Group 2 - Methylene blue (n=20) or Group 3 - Placebo (n=20)
5. 15 minutes after the initiation of CPB, the study drug will be administered intravenously through the central venous line by the anesthesia providers.
6. The study endpoints will be recorded from the anesthesia record above: MAP, CVP, CO, serum pH, pCO2 and lactate, vasopressor requirements, LVEF by TEE and end-tidal isoflurane dose at the following time points: 30 minutes after the induction of anesthesia (A), 15 minutes after the initiation of CPB just before the administration of study drug (pre-drug; time B), 30- and 60- minutes after the administration of study drug (post drug, times C and D), and 15-30 and 60-90 minutes after separation from CPB (post CPB, times E and F).
7. From the above measurements, calculated endpoints are derived: cardiac index calculated by CI=CO/body surface area (BSA), and systemic vascular resistance (SVR in dynes.s.cm-5) = (MAP-CVP)/CO x 800, and SVR index (SVRI) = (MAP-CVP)/CI x 800.
8. Follow-up will be carried out 24 hours after separation from CPB. Most patients are extubated in the intensive care unit at this time. The following data will be recorded: whether the patient has been extubated, vasopressor requirement, MAP and SVR, and adverse events at 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. 60 patients > 18 years of age
2. undergoing coronary artery bypass grafting (CABG) and/or valve surgery on cardiopulmonary bypass (CPB)
3. who have 2 or more preoperative risk factors for vasoplegia1-6:

   1. angiotensin-converting enzyme (ACE)-inhibitor, beta-blocker or amiodarone use within 24 hours of surgery
   2. anticipated CPB duration greater than 120minutes (combined CABG and valve procedure, >3 planned grafts, > 2 valve surgery)
   3. baseline left ventricular ejection fraction (LVEF) of less than 40%.

Exclusion Criteria:

1. Emergency surgery
2. Severe renal insufficiency (preoperative Cr > 1.8)
3. Severe hepatic disease (preoperative diagnosis of liver cirrhosis, or recent elevated liver function tests)
4. Pregnancy or women of childbearing potential
5. Known hypersensitivity to hydroxocobalamin or cyanocobalamin
6. Known hypersensitivity to methylene blue
7. Other known contraindications to methylene blue use: glucose-6-phosphate dehydrogenase (G6PD) deficiency, or ongoing selective serotonin reuptake inhibitor (SSRI), selective norepinephrine reuptake inhibitor (SNRI), tricyclic antidepressant (TCA) or monoamine inhibitor (MAOi) use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
ΔMAP (baseline to 30 min after CPB separation) in OH-CO and placebo groups. | From baseline to 30 minutes after successful separation from cardiopulmonary bypass (CPB)
  Our primary outcome measure is the change in MAP between one of the treatment (hydroxocobalamin) and placebo groups measured at 30 minutes post-CPB

SECONDARY OUTCOMES:
ΔMAP (baseline to 30 min after CPB separation) in OH-CO and MB groups. | From baseline to 30 minutes after successful separation from cardiopulmonary bypass (CPB)
  Our first secondary outcome measure is the change in MAP between the two treatment groups measured at 30 minutes post-CPB
ΔMAP between baseline and all time points (30 and 60 minutes after CPB initiation, and 30 and 60 minutes after CPB separation) between all 3 groups. | From baseline to all measured time points (30 and 60 minutes after CPB initiation, and 30 and 60 minutes after CPB separation).
  Our next secondary outcome measure is the change in MAP between all 3 groups at all measured time points.
ΔSVR (baseline to 30 min after CPB separation) in OH-CO and placebo groups. | From baseline to 30 minutes after successful separation from cardiopulmonary bypass (CPB)
  Change in SVR between one of the treatment (hydroxocobalamin) and placebo groups measured at 30 minutes post-CPB
ΔSVR (baseline to 30 min after CPB separation) in OH-CO and MB groups. | From baseline to 30 minutes after successful separation from cardiopulmonary bypass (CPB)
  Change in SVR between the two treatment groups measured at 30 minutes post-CPB
ΔSVR between baseline and all time points (30 and 60 minutes after CPB initiation, and 30 and 60 minutes after CPB separation) between all 3 groups. | From baseline to all measured time points (30 and 60 minutes after CPB initiation, and 30 and 60 minutes after CPB separation).
  Change in SVR between all 3 groups at all measured time points.
Differences in phenylephrine requirements during CPB between all 3 groups during CPB | At 30 and 60 minutes after initiation of CPB
  Phenylephrine dose in mcg/kg/min will be recorded from electronic medical record
Differences in Norepinephrine requirements during CPB between all 3 groups during and after CPB | At 30 and 60 minutes after initiation of CPB, and 30 and 60 minutes after separation from CPB
  Norepinephrine dose in mcg/kg/min will be recorded from electronic medical record
Differences in Vasopressin requirements during CPB between all 3 groups during and after CPB | At 30 and 60 minutes after initiation of CPB, and 30 and 60 minutes after separation from CPB
  Vasopressin dose in units/min will be recorded from electronic medical record

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No